CLINICAL TRIAL: NCT01989481
Title: Prospective Study of Risk Factors and Outcomes Following Total Knee Arthroplasty and Spinal Surgeon
Brief Title: Predicting the Outcome of Total Knee Arthroplasty and Spinal Surgeon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University Third Hospital (Other); Chinese PLA General Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Wei Tian, Director of Beijing Jishuitan Hospital, Beijing Jishuitan Hospital
Other Study IDs: 2012BAI10B02-OS
Record Dates: First submitted 2013-11-11; First posted 2013-11-21 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Osteoarthritis;; Intervertebral Disc Degeneration
MeSH Terms: conditions — Osteoarthritis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected from Peripheral Venous Blood； Tissues collected from the operation
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this observational study is to investigate the preoperative and operative factor of pain and functional outcome at one years following total knee arthroplasty and spinal surgeon.

ELIGIBILITY:
Inclusion Criteria:

1. The patients have been waiting for surgery for treatment of osteoarthritis or disc degeneration disease.
2. Must be between 18 and 65 years of age, of either sex.
3. Must demonstrate willingness to participate in the study by signing the written informed consent.

Exclusion Criteria:

1. Patients with Mandatory spondylitis, infections, neoplasms, inflammation, deformities, or previous surgery of spine or knee.
2. The patient is participating in an interventional clinical trial or has in an interventional clinical trial within 30 days prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients; Patients have been diagnosed with osteoarthritis or disc degeneration disease.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change of functional score over time in the patients after operation | 3, 6, 12 months after surgery

SECONDARY OUTCOMES:
Change of quality of life score over time in the patients after operation | 3, 6, 12 monthes after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tian, Doctor, Principal Investigator — Beijing Jishuitan Hospital
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China